CLINICAL TRIAL: NCT01386905
Title: A Study of the TransPyloric Shuttle™ (TPS™) for Weight Reduction in Obese Subjects (ENDObesity™ I Study)
Brief Title: A Study of the TransPyloric Shuttle™ (TPS™) for Weight Reduction in Obese Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BaroNova, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TPSS-I-0409-B
Record Dates: First submitted 2011-06-30; First posted 2011-07-01 (Estimated); Last update posted 2014-03-12 (Estimated); Status verified 2014-03

CONDITIONS: Obesity
Keywords: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: BAROnova™ TransPyloric Shuttle™ (TPS™) — Subjects will undergo an endoscopic procedure to deliver the TPS™ into the stomach. The TPS™ moves freely without any physical attachment or invasive anchoring to tissue to reduce gastric outflow.
  Other Names: ENDObesity I Study™; BAROnova™; TransPyloric Shuttle™; TPS™

SUMMARY:
The purpose of this study is to assess the feasibility of the TransPyloric Shuttle™ (TPS™) when used to treat obesity.

DETAILED DESCRIPTION:
The number of people who are overweight or obese has been steadily rising. In Australia, in 1980, 8.3% of the population was considered obese. By 2010, the Australian obesity rate had risen to 24.8%.

Weight loss significantly decreases early mortality as well as the development of new health-related conditions in obese subjects, and can improve many of the co-morbidities associated with obesity.

Therapies include drugs, surgery and treatment with medical devices, such as gastric banding and intragastric balloons. The TransPyloric Shuttle™ (TPS™) is a medical device that is endoscopically delivered and removed from the stomach. The TPS™ is designed to self-position across the pylorus and create an intermittent obstruction to outflow that may result in delayed gastric emptying. Slowing gastric emptying may enable an overall reduction in caloric intake by helping the subject feel full sooner (early satiation) and/or feel full longer (prolonged satiety/reduced hunger).

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects between the ages of 18 to 55.
2. BMI between 30 to 50 kg/m2. Subjects with BMI ≥ 35 to 50 kg/m2 inclusive, and subjects with a BMI of 30.0 to 34.9 kg/m2 are required to have one or more of the following obesity-related co-morbidities.

   1. Diabetes: controlled diabetic, and if on insulin, has been on the medication of less than two years.
   2. Sleep apnea: Apnea/hypopnea index or AHI > 30 events/hour.
   3. Hypertension: arterial blood pressure > 140 mmHg systolic or > 90 mmHg diastolic
   4. Osteoarthritis of the hip or knee.
   5. Gastro Esophageal Reflux Disease (GERD): Persistent reflux that occurs more than twice a week.
3. History of stable weight (defined as a < 10% change in excess weight) for one year prior to screening visit.
4. Female subjects of childbearing potential must have a negative urine pregnancy test and must agree to practice a medically acceptable form of birth control for the duration of their participation in the trial.
5. History of obesity for at least five years.
6. Subjects must be able to read and understand their native language at a level allowing the subject to understand and sign the informed consent prior to the performance of any study-specific procedure.
7. Lives within the drawing area of the hospital.
8. Willing and able to return for all study visits.

Exclusion Criteria:

1. Currently untreated thyroid and adrenal gland disease.
2. Females who are either pregnant or breastfeeding.
3. Insulin-dependent diabetic, where the subject has been on medication for more than two years.
4. Uncontrolled hypertension defined as systolic blood pressure > 160 mmHg or diastolic blood pressure > 95 mmHg.
5. Ischemic heart disease.
6. Previous stroke.
7. Previous myocardial infarct within 180 days of the study.
8. Prior history of bariatric surgery, such as gastric bypass, or any surgery that has altered the esophagus, stomach, or pylorus, and restrictive procedures such as the LAP-BAND® or equivalent.
9. Prior treatment with an intragastric balloon for the purpose of weight loss, where the balloon was removed less than 12 months prior to screening.
10. A structural abnormality in the esophagus, pharynx (such as a stricture), or pylorus (such as an incompetent pylorus).
11. Portal hypertension, cirrhosis, and/or varices.
12. Inflammatory disease, such as Crohn's disease, where the disease is affecting the stomach.
13. Acute abdominal infections.
14. Active gastric or duodenal ulcer.
15. A history of severe dyspepsia or gastric or duodenal ulcer disease.
16. After treatment for H. pylori, patient still tests positive for H. pylori.
17. Evidence of erosive esophagitis.
18. Subject with a hiatal hernia ≥ 2 cm.
19. Subjects with motility disorders of the GI tract such as esophageal motility disorders, gastroparesis diabeticorum, or intractable constipation.
20. Use of any prescription or over-the-counter weight loss medication, including herbal supplements, within three months of TPS device placement.
21. Subjects requiring continuous therapy with known ulcerogenic medication (e.g. aspirin, including 80 mg ASA or NSAIDs).
22. Subjects on anticoagulant therapy, such as those taking Coumadin, Warfarin, Heparin or Plavix.
23. Subjects unable to take a daily 40+ mg dose of Nexium or generic equivalent or 800+ mcg of Misoprostol or general equivalent.
24. Clinically significant abnormal laboratory values or EKG that make the subject a poor study candidate in the opinion of the investigator.
25. Subjects with autoimmune connective tissue disorders.
26. A history of cardiac arrhythmia or severe cardiac disease (NYHA Class III or IV).
27. Cannot walk at least 0.8 kilometers per day (10 minutes of continuous walking).
28. Subjects who have started on a prescribed concomitant medication regimen within the last three weeks, and/or whose concomitant medication regimen is expected to change during the course of the study, and where the Investigator determines the medication may affect the study outcome.
29. Treatment for drug abuse, alcohol abuse, or inpatient psychiatric treatment within the past year.
30. Any medical condition (including psychiatric disease) that would interfere with the interpretation of the study results, the conduct of the study, or would not be in the best interest of the subject.
31. A score of ≥ 10 on the Patient Health Questionnaire 9 (PHQ-9), indicating moderate depression.
32. Subjects who are in a dysfunctional relationship (e.g. an alcoholic spouse, the victim of sexual, verbal, or physical abuse, etc.).
33. Participation in a trial of an investigational drug or device within 30 days prior to Screening Visit or plans to enroll in an investigational drug or device trial at any time during this study.
34. Works for BAROnova or the study doctor or is directly-related to anyone that works for BAROnova or the study doctor.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2011-06; Primary Completion 2012-03 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Feasibility of the TransPyloric Shuttle™ System (TPS™) | Up to 6 months post-placement
  Preliminary evidence of the effectiveness of the TPS™ as determined by percent weight loss, excess BMI loss, and excess weight loss.

SECONDARY OUTCOMES:
Effect of the TransPyloric Shuttle™ (TPS™) on Patient Quality of Life | Up to 6 months post-placement
  Preliminary evidence of the effect of TPS™ on patient quality of life measured by lifestyle questionnaire 'Impact of Weight on Quality of Life-Lite' (IWQOL-Lite).
Safety of the TransPyloric Shuttle™ (TPS™) | Up to 6 months post-placement
  Preliminary evidence of TPS™ safety measured by device-related and procedure-related adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: George Marinos, MD, Principal Investigator — Gastric Balloon Australia
Locations (1):
- Gastric Balloon Australia (GBA), Bondi Junction, New South Wales, Australia

REFERENCES:
- [Background] Schols AM, Slangen J, Volovics L, Wouters EF. Weight loss is a reversible factor in the prognosis of chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 1998 Jun;157(6 Pt 1):1791-7. doi: 10.1164/ajrccm.157.6.9705017. PMID 9620907
- [Background] Sampalis JS, Liberman M, Auger S, Christou NV. The impact of weight reduction surgery on health-care costs in morbidly obese patients. Obes Surg. 2004 Aug;14(7):939-47. doi: 10.1381/0960892041719662. PMID 15329183
- [Result] http://www.oecd.org/document/16/0,2340,en_2649_34631_2085200_1_1_1_1,00.html